CLINICAL TRIAL: NCT00518531
Title: A Multicenter, Randomized, Cross-Over, Open-label Study to Evaluate the Adherence, Preference, and Satisfaction of Denosumab and Alendronate in Postmenopausal Women With Low Bone Mineral Density
Brief Title: Denosumab Adherence Preference Satisfaction Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20060232; DAPS
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Osteoporosis
Keywords: osteoporosis; low bone mineral density; alendronate; denosumab; adherence; preference; satisfaction; postmenopausal; women
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Personal Satisfaction | interventions — Alendronate; Denosumab

ARMS (2):
- Treatment Sequence B (Other): When a subject meets all eligibility criteria and signs the informed consent, they will be randomized in a 1:1 allocation to one of the two treatment Sequences. Subjects randomized to treatment sequence B will receive 70 mg oral alendronate QW for 1-year (Treatment period 1) followed by denosumab 60 mg Q6M SC for 1 year (Treatment Period 2).
  Interventions: Drug: alendronate; Drug: denosumab
- Treatment Sequence A (Other): When a subject meets all eligibility criteria and signs the informed consent, they will be randomized in a 1:1 allocation to one of the two treatment sequences. Subjects randomized to treatment sequence A will receive 60 mg denosumab Q6M SC for 1-year (Treatment period 1) followed by oral alendronate 70 mg QW for 1 year (Treatment period 2).
  Interventions: Drug: alendronate; Drug: denosumab

INTERVENTIONS:
Drug: alendronate — Subjects will take 70 mg QW of oral alendronate for 1 year. If a subject is randomized to Treatment Sequence A they will receive alendronate for 1 year in Treatment Period 2. If a subject is randomized to Treatment Sequence B they will receive alendronate for 1 year in Treatment Period 1.
Drug: denosumab — Subjects will receive 60 mg of denosumab Q6M SC for 1 year. If a subject is randomized to Treatment Sequence A they will receive denosumab for 1 year in Treatment Period 2. If a subject is randomized to Treatment Sequence B they will receive denosumab for 1 year in Treatment Period 1.

SUMMARY:
The primary objective is to evaluate the adherence of subjects to subcutaneous (SC) 60 mg denosumab every 6 months (Q6M) treatment compared to oral 70 mg alendronate once a week (QW) treatment at the end of treatment period 1 (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women based on medical history
* > or = 55 years of age at the start of screening
* Screening bone mineral density (BMD) values (g/cm²), at the lumbar spine OR femoral neck OR total hip that occur within the specified ranges based on the particular scanner that is used. At least 2 lumbar vertebrae must be evaluable by Dual X-ray Absorptiometry (DXA), or at least one hip must be evaluable by DXA
* Provide written informed consent before any study specific procedure is performed.

Exclusion Criteria:

* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Hyper- or hypothyroidism; however, stable subjects, in the investigator's opinion, on thyroid hormone replacement therapy are allowed
* Current hyper- or hypoparathyroidism
* Current hypo- or hyper calcemia based on the central laboratory reference ranges for albumin-adjusted serum calcium
* Rheumatoid arthritis, Paget's disease, Cushing's disease, hyperprolactinemia, or cirrhosis of the liver
* Any metabolic bone disease, e.g. osteomalacia or osteogenesis imperfecta, which may interfere with the interpretation of the findings
* Any symptomatic vertebral fracture within 3 months prior to screening
* Previous participation in clinical trials with denosumab
* Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (<49.9 nmol/L)]
* Contraindicated to alendronate therapy; contraindications for alendronate therapy include:

  1. Abnormalities of the esophagus, which delay esophageal emptying such as stricture or achalasia.
  2. Inability to stand or sit upright for at least 30 minutes.
  3. Hypersensitivity to alendronate (ALN) or other constituents of ALN tablets.
* Any known prior bisphosphonate use
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trail (s), or subject is receiving other investigational agent(s).

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2010-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Freemantle N, Satram-Hoang S, Tang ET, Kaur P, Macarios D, Siddhanti S, Borenstein J, Kendler DL; DAPS Investigators. Final results of the DAPS (Denosumab Adherence Preference Satisfaction) study: a 24-month, randomized, crossover comparison with alendronate in postmenopausal women. Osteoporos Int. 2012 Jan;23(1):317-26. doi: 10.1007/s00198-011-1780-1. Epub 2011 Sep 17. PMID 21927922
- [Background] Kendler DL, Macarios D, Lillestol MJ, Moffett A, Satram-Hoang S, Huang J, Kaur P, Tang ET, Wagman RB, Horne R. Influence of patient perceptions and preferences for osteoporosis medication on adherence behavior in the Denosumab Adherence Preference Satisfaction study. Menopause. 2014 Jan;21(1):25-32. doi: 10.1097/GME.0b013e31828f5e5d. PMID 23676636
- [Background] Kendler DL, McClung MR, Freemantle N, Lillestol M, Moffett AH, Borenstein J, Satram-Hoang S, Yang YC, Kaur P, Macarios D, Siddhanti S; DAPS Investigators. Adherence, preference, and satisfaction of postmenopausal women taking denosumab or alendronate. Osteoporos Int. 2011 Jun;22(6):1725-35. doi: 10.1007/s00198-010-1378-z. Epub 2010 Sep 9. PMID 20827547
- [Derived] Kendler D, Chines A, Clark P, Ebeling PR, McClung M, Rhee Y, Huang S, Stad RK. Bone Mineral Density After Transitioning From Denosumab to Alendronate. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e255-64. doi: 10.1210/clinem/dgz095. PMID 31665314
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 03-Oct-07, last subject enrolled 25-Jun-08; First subject crossovered 22-May-08, last subject crossovered 25-Jun-09;
Groups:
- Alendronate in Period 1 Then Denosumab in Period 2: Alendronate 70 mg orally once a week (QW) for 1 year (treatment period 1) followed by Denosumab 60 mg subcutaneously every 6 months for 1 year (treatment period 2).
- Denosumab in Period 1 Then Alendronate in Period 2: Denosumab 60 mg subcutaneously every 6 months for 1 year (treatment period 1) followed by Alendronate 70 mg orally once a week for 1 year (treatment period 2).
Period: Treatment Period 1
Arm/Group | Alendronate in Period 1 Then Denosumab in Period 2 | Denosumab in Period 1 Then Alendronate in Period 2
Started | 124 | 126
Received Treatment | 119 | 124
Completed | 106 | 114 (Participants who completed Treatment Period 1 may choose not to start Treatment Period 2)
Not Completed | 18 | 12
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 5 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Early crossover | 1 | 3
Period: Treatment Period 2
Arm/Group | Alendronate in Period 1 Then Denosumab in Period 2 | Denosumab in Period 1 Then Alendronate in Period 2
Started | 106 | 115 (Participants can start Treatment Period 2 without completing Treatment Period 1.)
Received Treatment | 106 | 110
Completed | 103 | 95
Not Completed | 3 | 20
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Complete out of scheduled visit window | 1 | 2
Not completed — Adverse Event | 1 | 7
Not completed — Protocol-specified criteria | 0 | 1
Not completed — Non-compliance | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Alendronate in Period 1 Then Denosumab in Period 2: Alendronate 70 mg orally once a week for 1 year (treatment period 1) followed by Denosumab 60 mg subcutaneously every 6 months for 1 year (treatment period 2).
- Total: Total of all reporting groups
Arm/Group | Alendronate in Period 1 Then Denosumab in Period 2 | Denosumab in Period 1 Then Alendronate in Period 2 | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (7.7) | 65.1 (7.6) | 65.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 126 | 250
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 119 | 115 | 234
  Black or African American | 2 | 2 | 4
  Hispanic or Latino | 1 | 6 | 7
  Asian | 1 | 3 | 4
  Japanese | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Treatment in the First Treatment Period
Description: A participant was considered adherent to denosumab treatment if the participant: - received 2 denosumab injections (overall treatment compliance); - took each injection 6 months (± 4 weeks) apart (treatment compliance over time); - completed the relevant treatment period (treatment persistence). A participant was considered adherent to alendronate treatment if the participant: - took ≥ 80% QW tablets (overall treatment compliance); - took at least 2 tablets in the last month and completed the relevant treatment period (treatment persistence). Participants who did not meet all criteria for their assigned treatment were deemed non-adherent to treatment.
Time Frame: Treatment period 1 (Month 1 to Month 12)
Population: The full analysis set (FAS) includes all participants who were randomized.
Measure: Number; unit: Participants
Groups:
- Alendronate: Participants received alendronate 70 mg orally once a week for 1 year.
- Denosumab: Participants received denosumab 60 mg subcutaneously every 6 months for 1 year.
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 124 | 126
Participants
  Yes | 95 | 111
  No | 29 | 15
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p = 0.0259, Cochran-Mantel-Haenszel — All statistical hypothesis tests were conducted at the 0.05 significance level. No adjustment was employed for multiple comparisons; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 10.5, 95% CI 2-sided [1.3 to 19.7] — Positive values for absolute risk reduction favor denosumab

2. Secondary Outcome: Adherence With Treatment in the Second Treatment Period
Description: A participant was considered adherent to denosumab treatment if the participant: - received 2 denosumab injections (overall treatment compliance); - took each injection 6 months (± 4 weeks) apart (treatment compliance over time); - completed the relevant treatment period (treatment persistence). A participant was considered adherent to alendronate treatment if the participant: - took ≥ 80% QW tablets (overall treatment compliance); - took at least 2 tablets in the last month and completed the relevant treatment period (treatment persistence). Participants who did not meet all criteria for their assigned treatment were deemed nonadherent to treatment.
Time Frame: Treatment period 2 (Months 13 to 24)
Population: The cross-over analysis set includes all participants who crossed over to their treatment period 2 treatment.
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 106
Participants
  Yes | 73 | 98
  No | 42 | 8
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 30.9, 95% CI 2-sided [20.6 to 41.3] — Positive values for absolute risk reduction favor denosumab

3. Secondary Outcome: Compliance With Treatment in the First Treatment Period
Description: Participants were considered compliant to denosumab treatment if they received 2 denosumab injections (overall treatment compliance) and if they took each injection 6 months (± 4 weeks) apart (treatment compliance over time). Participants were considered compliant to alendronate treatment if they took ≥ 80% QW tablets (overall treatment compliance).
Time Frame: Treatment period 1 (Month 1 to Month 12)
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 124 | 126
Participants
  Yes | 97 | 114
  No | 27 | 12
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p = 0.0138, Cochran-Mantel-Haenszel; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 11.00, 95% CI 2-sided [2.2 to 19.7] — Positive values for absolute risk reduction favor denosumab

4. Secondary Outcome: Compliance With Treatment in the Second Treatment Period
Description: as for outcome 3
Time Frame: Treatment period 2 (Month 13 to Month 24)
Population: Crossover set
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 106
Participants
  Yes | 78 | 99
  No | 37 | 7
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 27.7, 95% CI 2-sided [17.6 to 37.7] — Positive values for absolute risk reduction favor denosumab

5. Secondary Outcome: Persistence With Treatment in the First Treatment Period
Description: Denosumab-treated participants were considered persistent to treatment if they completed the relevant treatment period and alendronate-treated participants were considered persistent to treatment if they completed the relevant treatment period and took at least 2 tablets in the last month of the treatment period.
Time Frame: Treatment period 1 (Month 1 to Month 12)
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 124 | 126
Participants
  Yes | 99 | 114
  No | 25 | 12
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p = 0.0291, Cochran-Mantel-Haenszel; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 9.8, 95% CI 2-sided [1.1 to 18.5] — Positive values for absolute risk reduction favor denosumab

6. Secondary Outcome: Persistence With Treatment in the Second Treatment Period
Description: as for outcome 5
Time Frame: Treatment period 2 (Month 13 to Month 24)
Population: Crossover set
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 106
Participants
  Yes | 82 | 103
  No | 33 | 3
Statistical Analysis 1: Comparison: Alendronate vs Denosumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by center and prior osteoporotic fracture; Risk Difference (RD) = 27.4, 95% CI 2-sided [18.1 to 36.7] — Positive values for absolute risk reduction favor denosumab

7. Secondary Outcome: Time to Non-adherence to Alendronate Treatment in the First Treatment Period
Description: Time to treatment non-adherence for alendronate is defined for each treatment period as the time to treatment non-compliance or time to treatment non-persistence, whichever occurs earliest, for participants with uncensored values. Participants who had both censored time to non-compliance and censored time to non-persistence values were censored in the analysis at the end of treatment period visit.
Time Frame: Treatment Period 1 (Month 1 to Month 12)
Population: Full analysis set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 124
weeks | 43.29 (1.46)

8. Secondary Outcome: Time to Non-adherence to Alendronate Treatment in the Second Treatment Period
Description: as for outcome 7
Time Frame: Treatment Period 2 (Month 13 to Month 24)
Population: Crossover set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 115
weeks | 39.45 (1.89)

9. Secondary Outcome: Time to Non-compliance to Alendronate Treatment in the First Treatment Period
Description: Time to treatment non-compliance for alendronate is based on the percent of QW tablets taken and is defined for each treatment period as the first week since Study Day 1 of the treatment period to the week where the percent of QW tablets taken falls below the threshold of ≥ 80% and where the participant can not reach this threshold again during the treatment period.
Time Frame: Treatment period 1 (Month 1 to Month 12)
Population: Full analysis set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 124
weeks | 43.75 (1.42)

10. Secondary Outcome: Time to Non-compliance to Alendronate Treatment in the Second Treatment Period
Description: as for outcome 9
Time Frame: Treatment period 2 (Month 13 to Month 24)
Population: crossover set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 115
weeks | 39.97 (1.87)

11. Secondary Outcome: Time to Non-persistence to Alendronate Treatment in the First Treatment Period
Description: Time to non-persistence for alendronate is defined for each treatment period as the first time <2 tablets were taken in a rolling 4-week time period (e.g. study weeks 1-4, 2-5, 3-6 etc) and where the participant never reaches this threshold again during the treatment period. Tablet intake was tracked using a Medication Event Monitoring System.
Time Frame: Treatment period 1 (Month 1 to Month 12)
Population: Full analysis set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 124
weeks | 44.59 (1.35)

12. Secondary Outcome: Time to Non-persistence to Alendronate Treatment in the Second Treatment Period
Description: as for outcome 11
Time Frame: Treatment period 2 (Month 13 to Month 24)
Population: Crossover set
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Alendronate
Number analyzed (Participants) | 115
weeks | 42.76 (1.69)

13. Secondary Outcome: Overall Satisfaction to Study Treatment
Description: Participant satisfaction with their treatment was assessed using question 7 (ie, "Please rate your satisfaction with the weekly pill on the following: frequency of administration; mode of administration [taking a pill]; convenience; overall satisfaction") and question 8 (ie, "Please rate your satisfaction with the six month injection on the following: frequency of administration; mode of administration [receiving an injection]; convenience; overall satisfaction") from the Preference Satisfaction Questionnaire (PSQ) at the end of each treatment period. The PSQ is a 34 item, self-report questionnaire of participants' preference and satisfaction for each of the two study treatments. Possible answers include: "Not at all Satisfied", "A Little Satisfied", "Moderately Satisfied", "Quite Satisfied", and "Very Satisfied".
Time Frame: End of treatment period 1 (Month 12)
Population: The Patient Reported Outcomes (PRO) analysis set for each independent treatment period included patients in the FAS who received at least one dose of study drug and had at least one post-baseline assessment in the relevant treatment period. Analysis population includes patients with observed data for ≥1 question in the questionnaire.
Measure: Number; unit: Participants
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 114 | 121
Participants
  Not at all satisfied | 3 | 3
  A little satisfied | 1 | 3
  Moderately satisfied | 17 | 2
  Quite satisfied | 34 | 18
  Very satisfied | 59 | 95

14. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ): Necessity Score
Description: The BMQ is a 22- item self-reported questionnaire specific to osteoporosis that measures beliefs about the weekly pill or every 6 months injection. The BMQ consists of 3 subscales measuring beliefs about the necessity of the medication for controlling osteoporosis, concern with the adverse consequences of taking the medication, and preference for one medication over the other.
  Participants' beliefs about the necessity of the prescribed medication to treat osteoporosis were based on the average of 5 items from the BMQ that form the necessity score. The necessity score ranges from 1 to 5, with higher scores indicating stronger beliefs about the necessity of the prescribed medication for controlling osteoporosis.
Time Frame: Baseline, Month 6, Month 12, Month 18 and Month 24
Population: Participants in the PRO analysis set with observed data; "n" indicates the number of patients with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 121
scores on a scale
  Baseline (n=104, 117) | 3.32 (0.52) | 3.26 (0.48)
  Month 6 (n=106, 114) | 3.14 (0.53) | 3.31 (0.60)
  Month 12 (n=103, 95) | 3.21 (0.51) | 3.17 (0.52)
  Month 18 (n=98, 98) | 3.20 (0.53) | 3.28 (0.55)
  Month 24 (n=91, 100) | 3.21 (0.62) | 3.22 (0.58)

15. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ) Concern Score
Description: The BMQ is a 22- item self-reported questionnaire specific to osteoporosis that measures beliefs about the weekly pill or every 6 months injection. The BMQ consists of 3 subscales measuring beliefs about the necessity of the medication for controlling osteoporosis, concern with the adverse consequences of taking the medication, and preference for one medication over the other. Participants' concern about the adverse consequences of taking the medication for controlling osteoporosis was based on the average of 10 items from the BMQ that form the concern score. The concern score ranges from 1 to 5, with higher scores indicating stronger concerns about the adverse consequences of taking the prescribed medication for controlling osteoporosis.
Time Frame: Baseline and Month 6, Month 12, Month 18, and Month 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 121
scores on a scale
  Baseline (n=104, 117) | 2.33 (0.48) | 2.43 (0.46)
  Month 6 (n=106, 114) | 2.22 (0.51) | 2.12 (0.51)
  Month 12 (n=103, 95) | 2.57 (0.48) | 2.51 (0.50)
  Month 18 (n=98, 98) | 2.43 (0.58) | 2.24 (0.49)
  Month 24 (n=91, 100) | 2.39 (0.58) | 2.18 (0.51)

16. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ) Preference Score
Description: The BMQ is a 22- item self-reported questionnaire specific to osteoporosis that measures beliefs about the weekly pill or every 6 months injection. The BMQ consists of 3 subscales measuring beliefs about the necessity of the medication for controlling osteoporosis, concern with the adverse consequences of taking the medication, and preference for one medication over the other. The BMQ preference score, which measures a participant's overall evaluation of a medication, is based on the average of 7 items in the BMQ. The preference score ranges from 1 to 5, with higher scores indicating stronger preference for one medication over the other.
Time Frame: Baseline and Month 6, Month 12, Month 18, and Month 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Alendronate | Denosumab
Number analyzed (Participants) | 115 | 121
scores on a scale
  Baseline (n=104, 117) | 2.97 (0.40) | 3.47 (0.43)
  Month 6 (n=106, 114) | 3.01 (0.53) | 3.72 (0.47)
  Month 12 (n=103, 95) | 2.62 (0.50) | 3.43 (0.45)
  Month 18 (n=98, 98) | 2.55 (0.56) | 3.77 (0.47)
  Month 24 (n=91, 100) | 2.57 (0.65) | 3.80 (0.52)

17. Secondary Outcome: Medication Adherence Rating Scale (MARS) to Alendronate in the First Treatment Period
Description: The MARs questionnaire is a validated, self-reported instrument for assessing treatment adherence. Participants report how often they engage in each of 5 aspects of non-adherent behavior (forgetting to take a dose, changing the dose, stop taking them for a while, deciding to not take a dose, or taking less than instructed). Scores are summed over the 5 items, the total score ranges from 5 to 25 with higher scores indicating greater self-reported adherence. The MARS was collected at the month 6 and month 12 visits of each treatment period only for those participants receiving oral alendronate during that period.
Time Frame: Month 6, Month 12 (treatment period 1)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Alendronate
Number analyzed (Participants) | 115
scores on a scale
  Month 6 (n=109) | 24.3 (1.1)
  Month 12 (n= 100) | 24.4 (1.4)

18. Secondary Outcome: Medication Adherence Rating Scale (MARS) to Alendronate in the Second Treatment Period
Description: as for outcome 17
Time Frame: Month 18, Month 24 (treatment period 2)
Population: Participants in the PRO analysis set with at least one post-baseline assessment in both periods and with observed data; "n" indicates the number of patients with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Alendronate
Number analyzed (Participants) | 100
scores on a scale
  Treatment period 2 Month 6 (n=98) | 23.4 (2.0)
  Treatment period 2 Month 12 (n= 90) | 23.8 (1.4)

ADVERSE EVENTS:
Time Frame: 24 months
Description: In Treatment Period 1, one participant received both treatments and is counted in the denosumab group for safety analyses.
  The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Groups:
- Treatment Period 1: Alendronate: Participants received alendronate 70 mg orally once a week in year 1.
- Treatment Period 1: Denosumab: Participants received denosumab 60 mg subcutaneously every 6 months in year 1.
- Treatment Period 2: Alendronate: Participants who received denosumab 60 mg subcutaneously every 6 months in year 1 then received alendronate 70 mg orally once a week in year 2.
- Treatment Period 2: Denosumab: Participants who received alendronate 70 mg orally once a week in year 1 then received denosumab 60 mg subcutaneously every 6 months in year 2.
Arm/Group | Treatment Period 1: Alendronate | Treatment Period 1: Denosumab | Treatment Period 2: Alendronate | Treatment Period 2: Denosumab
Serious Adverse Events (participants affected / at risk) | 5/118 | 4/125 | 4/110 | 4/106
Other Adverse Events (participants affected / at risk) | 24/118 | 31/125 | 21/110 | 13/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: Alendronate (N=118) | Treatment Period 1: Denosumab (N=125) | Treatment Period 2: Alendronate (N=110) | Treatment Period 2: Denosumab (N=106)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pelvic mass (General disorders) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: Alendronate (N=118) | Treatment Period 1: Denosumab (N=125) | Treatment Period 2: Alendronate (N=110) | Treatment Period 2: Denosumab (N=106)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11 | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 9 | 4 | 5
Headache (Nervous system disorders) | 7 | 4 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.